

# RETROSPECTIVE OBSERVATIONAL COHORT STUDY SYMBOL CUP 2

#### SYMCOR-2

Version N°1.0- Date: 16-APR-2018

| Investigator | Dr. Gilles ESTOUR |
|--------------------------|--------------------------------------------------|
| Sponsor | DEDIENNE SANTE SAS represented by Ludovic TOLEDO |
| Methodology & Biometrics | Prof. Dr. Frédéric DAOUD |

This document is the exclusive property of the sponsor. It may not be copied, reproduced or communicated, in whole or in part, without written authorization.



# **KEY STAKEHOLDERS**

| Sponsor | DEDIENNE SANTE S.A.S. |
|---------------------------|-------------------------------------------------|
| | SIRET: 339 138 638 00053 |
| | 217, rue Charles Nungesser, 34130 Mauguio |
| | Represented by TOLEDO Ludovic, General Director |
| | Phone: 04 67 99 81 11 |
| | Mail: l.toledo@menix.fr |
| Investigator | Dr. Gilles ESTOUR |
| | RPPS 10004039441 |
| | Orthopedic Surgeon |
| | MEDIPOLE DE SAVOIE |
| | Avenue des Massettes |
| | 73190 Challes-les-Eaux |
| | Phone: 04 79 26 81 17 |
| | Mail: gillestour@yahoo.com |
| Methodology and data | Dr. Frédéric DAOUD |
| management: place of data | RPPS 10000548973 |
| processing | Epidemiologist, biostatistician. |
| | MEDEXTENS SARL |
| | 75 rue de Lourmel, 75015 Paris |
| | Phone: 06 03 00 68 98 |
| | Mail: fcdaoud@medextens.com |



# PROTOCOL UPDATE HISTORY

| VERSION | DATE | REASON FOR UPDATE |
|---------|------------|-------------------|
| 1.0 | 16/04/2018 | Final version |



| 1. | SUMMARY ( | OF THE STUDY | 6 |
|---|---|---|---|
| 2. | STUDY RAT | IONALE / SCIENTIFIC JUSTIFICATION | 7 |
| | 2.1. | CURRENT KNOWLEDGE OF THE PATHOLOGY | 7 |
| | 2.2. | STATE OF KNOWLEDGE ON THE DEVICES UNDER EVALUATION | 10 |
| | 2.3. | STUDY HYPOTHESES AND EXPECTED RESULTS | 11 |
| 3. | STUDY OBJI | ECTIVES AND ENDPOINTS | 11 |
| | 3.1. | MAIN OBJECTIVE | 11 |
| | 3.2. | PRIMARY ENDPOINT | 12 |
| | 3.3. | SECONDARY OBJECTIVE | 12 |
| | 3.4. | SECONDARY ENDPOINTS | 12 |
| 4. | DESCRIPTION | ON OF THE STUDY | 12 |
| | 4.1. | DESCRIPTION OF MEASURES TAKEN TO REDUCE AND AVOID BIAS | 12 |
| 5. | STUDY FEAS | SABILITY | 13 |
| 6. | REALISATIO | ON PRATIQUE DU PROTOCOLE. | 13 |
| | 6.1. | DEROULEMENT DES VISITES LIEES A L'ETUDE | 13 |
| | 6.2. | SUMMARY OF PATIENT FOLLOW-UP | 14 |
| | 6.3. | DESCRIPTION OF THE GENERAL LOGISTICAL ORGANIZATION OF THE STUDY | 14 |
| | 6.4. | BIOLOGICAL SAMPLES AND ANALYSES | 14 |
| 7. | ELIGIBILIT | Y CRITERIA | 14 |
| | 7.1. | INCLUSION CRITERIA | 14 |
| | 7.2. | Non-inclusion criteria | 14 |
| | 7.3. | RECRUITMENT PROCEDURES | 15 |
| 8. | RULES FOR | STOPPING THE STUDY | 15 |
| | 8.1. | TERMINATION OF THE STUDY BY THE SPONSOR | 15 |
| | 8.2. | TERMINATION OF THE STUDY BY THE INVESTIGATOR | 15 |
| 9. | DATA COLL | ECTED | 15 |
| 10. | STATISTICA | AL CONSIDERATIONS | 15 |
| | 10.1. | NUMBER OF SUBJECTS TO BE INCLUDED | 15 |
| | 10.2. | DATA ANALYSIS – GENERAL INFORMATION: DESCRIPTIVE APPROACH | 15 |
| | 10.3. | MAIN ANALYSIS | 16 |
| | 10.4. | SECONDARY ANALYSES | 16 |
| | 10.5. | SAMPLING FRAME | 16 |
| | 10.6. | METHOD FOR TAKING INTO ACCOUNT MISSING, UNUSED OR INVALID DATA | 16 |
| | 10.7. | PERSON RESPONSIBLE FOR THE ANALYSIS | 16 |



| 11. | ACCESS RIGI | HTS TO SOURCE DATA AND DOCUMENTS | 17 |
|---|---|---|---|
| 1 | 1.1. | DATA ACCESS | 17 |
| 1 | 1.2. | SOURCE DATA | 17 |
| 1 | 1.3. | DATA PRIVACY | 17 |
| 12. | ETHICAL CO | NSIDERATIONS | 18 |
| 1 | 2.1. | INDEPENDENT ETHICS COMMITTEE | 18 |
| 1 | 2.2. | PATIENT INFORMATION | 18 |
| 1 | 2.3. | SUPPORT FOR STUDY | 18 |
| 13. | DATA PROC | ESSING AND STORAGE OF DOCUMENTS AND DATA RELATING T | го тне |
| STU | DY | | 19 |
| 1 | 3.1. | DATA ENTRY AND PROCESSING | 19 |
| 1 | 3.2. | CNIL | 19 |
| 1 | 3.3. | ARCHIVING | 19 |
| 14. | COMMUNICA | ATION – PUBLICATION RULES | 19 |
| 15. | INVESTIGAT | OR CONTRACT | 20 |
| 16. | LIST OF ANN | EXES | 20 |
| 17. | ASSOCIATED | DOCUMENTS | 20 |
| 18. | BIBLIOGRAP | РНУ | 37 |

# 1. SUMMARY OF THE STUDY

| TITLE | Retrospective Observational Cohort Study SYMBOL CUP 2 |
|---|---|
| SHORT TITLE | SYMCOR-2 |
| INVESTIGATOR | Dr. Gilles ESTOUR |
| SPONSOR | DEDIENNE SANTE S.A.S. |
| JUSTIFICATION / CONTEXT | Documentation of the clinical efficacy and safety of SYMBOL CUP DMR HA and SYMBOL CUP DM CEM dual mobility acetabular implants. |
| METHODOLOGY | Retrospective observational cohort study |
| MAIN OBJECTIVE | Estimate the safety of these implants under normal conditions of use |
| PRIMARY ENDPOINT | Implant survival rate at 2-year follow-up |
| SECONDARY OBJECTIVE | Estimate the efficacy of these implants under normal conditions of use |
| SECONDARY ENDPOINTS | - Safety: Intra and extra-prosthetic dislocation rates |
| | - Safety: Incidence of other adverse events |
| | - Effectiveness: Harris Hip Score (HHS) |
| | - Effectiveness: Devane classification |
| | - Effectiveness: Charnley classification |
| | - Any patient operated by Dr. Estour who has undergone hip |
| INCLUSION CRITERIA | replacement surgery with SYMBOL CUP DMR HA or SYMBOL |
| | CUP CEM acetabular implant. |
| | - Patient having reach 2-year follow-up on March 01, 2018 |
| NON-INCLUSION | - Explicit refusal by the patient to allow data describing his |
| CRITERIA | pathology and treatment to be included in this study. |
| | - Minor patients or patients under guardianship. |



| | Detroprocing collection of clinical data: |
|---|---|
| | Retrospective collection of clinical data: |
| | - Recorded in the orthopedic surgery department's patient files, |
| | from the patient's pre-surgical assessment to the latest news at 2- |
| Drop a now process | year follow-up. |
| RESEARCH PROCESS | - Obtained by telephone interview for data up to 2-year follow-up, |
| | if the medical file does not provide all the source information. The |
| | telephone interview will be carried out by the investigator (or his |
| | secretariat) or by a clinical research associate delegated by the |
| | sponsor and approved by the investigator. |
| NUMBER OF SUBJECTS | Minimum total number of subjects: n=20 |
| | Minimum total number of subjects: n=20 |
| PLANNED NUMBER OF | |
| CENTERS | Single-center, single-investigator study |
| | CPP notice: N.A. |
| | CEREES notice: N.A. |
| | CNIL receipt: 2176595 |
| PROVISIONAL STUDY | Start of the study: As soon as CNIL receipt is received. |
| TIMETABLE | Duration of inclusion period/data collection: N.A. given retrospective |
| | nature |
| | Duration of participation of each subject: N.A. given retrospective nature |
| | Anticipated end of study: N.A. given retrospective nature |
| | End-of-study report: Within 30 days of start of study |
| | - Descriptive statistics: preoperative, operative, postoperative |
| STATISTICAL DATA | - Tabulation of adverse events |
| ANALYSIS | - Kaplan-Meier analysis of implant survival |
| | - Comparison tests of preoperative versus 1-year and 2-year |
| | postoperative efficacy scores. |
| | I . |

# 2. STUDY RATIONALE / SCIENTIFIC JUSTIFICATION

# 2.1. <u>CURRENT KNOWLEDGE OF THE PATHOLOGY</u>

Hip replacement is the last therapeutic resort for symptomatic coxopathies, the incidence of which is estimated at over 85,000 patients per year, if hip replacement is considered as an indicator of this



pathology, according to data from the Programme de Médicalisation des Systèmes d'Information (PMSI).

In the report of 2014, the Haute Autorité de Santé<sup>i</sup>, recommends the use of dual-mobility acetabular implants:

- In first-line arthroplasties in patients with a very high risk of dislocation (severe neurological impairment, neuropsychiatric disorders, addiction, and major neuromuscular failures),
- And revision arthroplasties in case of iterative dislocation and in patients at high rik of dislocation,
- Depending on the clinical situation, press-fit fixation is the preferred method of fixation for the metal-back dual mobility acetabular cups, when the bone bed is of good quality.

In current practice, dual-mobility acetabular implants with cemented fixation in a cross shell, or with cortical screws and peg, are chosen when damage to the bed bone is extensive and does not allow direct press-fit implantation. This is particularly the case in revision surgery.

SYMBOL CUP DMR HA acetabular implants comprise metal-back cup with cortical screw fixation and peg fixation and the same DUAL MOBILITY PE LINER dual-mobility polyethylene insert as in all acetabular implants in the SYMBOL CUP DM range (Table 1, Figure 1).

Table 1: SYMBOL CUP DMR HA with cortical screw and pegs: technical specifications

| | RANGE (Manufacturer) | SYMBOL CUP<br>DMR HA<br>(Dedienne<br>Santé) | Also sold under the brand names: GYRACUP Ultimate (AESCULAP), DS Evolution (MATHYS Ltd.) | |
|---|---|---|---|---|
| | Model | Symbol Cup DMR | НА | |
| | Diameter range | 44 to 68mm | | |
| Cups | Metal-back material | Co-Cr (ISO 5832-4) | | |
| Оцро | Coating | | Ti +HAP (ISO 13779-2) | |
| | Fixation | * Press-Fit +<br>Tripod | * 2 pegs through holes in cups | * 1 cortical screw in the flange |
| | Model | Dual Mobility PE Liner | | |
| Material | | polyethylene ISO 5834-2 UHMWPE | | |
| Liners | Diameter range | | 44 to 68mm | |
| Range of diameters for corresponding femoral heads 22,2mm or 28mm | | | | |



Figure 1 Photos of SYMBOL CUP DMR HA and PE LINER medical devices.



SYMBOL CUP DM CEM acetabular implants comprise a metal-back cup designed to be cemented to the surrounding bone, and the same DUAL MOBILITY PE LINER dual-mobility polyethylene insert as in all acetabular implants in the SYMBOL CUP DM range (Table 2, Figure 2).

Table 2: SYMBOL CUP DM CEM to be cemented: technical specifications.

| | RANGE (Manufacturer) | SYMBOL CUP DM<br>CEM (Dedienne<br>Santé) | Also sold under the brand names:<br>GYRACUP E (AESCULAP), DS<br>Evolution (MATHYS Ltd.) |
|---|---|---|---|
| | Model | Symbol Cup DM CEM | Л |
| | Diameter range | 44 to 68mm | |
| Cups | Metal-back material | Co-Cr (ISO 5832-4) | |
| | Coating | N.A | |
| | Fixation | Cement | |
| | Model | Dual Mobility PE Line | r |
| | Material | polyethylene ISO 583 | 34-2 UHMWPE |
| Liners | Diameter range | 44 to 68 mm | |
| | Range of diameters for corresponding femoral heads | 22,2mm or 28mm | |

Figure 2 Photos of SYMBOL CUP DM CEM and PE LINER medical devices.





## 2.2. STATE OF KNOWLEDGE ON THE DEVICES UNDER EVALUATION

SYMBOL CUP DMR HA and SYMBOL CUP DM CEM are class III implantable devices according to rule N°20 of the decree of April 20, 2006, laying down the rules for the classification of medical devices (transposition of Annex IX of directive 93/42/EEC and Directive 2005/50/EC).

These implants have been introduced on the market in France and elsewhere in Europe since the EC declaration of conformity of April 09, 2014<sup>ii</sup>. Conformity in based in particular on:

- Certificate N°27262 of device design examination according to Annex II section 4 if Directive 93/42/EEC issued by the Notified Body LNE/G-MED N°0459, updated by revision 5 dated September 01, 2015.<sup>iii</sup>
- The clinical evaluation « Cotyles de hanche, double mobilité, SYMBOL CUP DM » dated 28/11/2013 performed by Dedienne Santé, updated on 28/11/2014.iv
- And the validation of the clinical evaluation report by the Notified Body LNE/G-MED.<sup>v</sup>

The clinical evaluation of SYMBOL CUP DMR HA and SYMBOL CUP DM CEM as part as CE conformity is based on a literature review of equivalent products, with no data specific to these products. Nevertheless, the CE mark has authorized SYMBOL CUP DMR HA to be reimbursed by the French health insurance, under the Liste des Produits et Prestations Remboursables, under generic code 3168042 (reconstruction cup, modular, metal-back, without insert, uncemented) and SYMBOL CUP DM CEM under generic code 3150450 (standard cup, modular, metal-back, without insert, cemented). In both cases, the insert was covered under generic code 3161130 (solid polymer insert). The patients identified for this retrospective study benefited from reimbursement of the implant according to these generic codes.

Given the relatively recent market introduction of SYMBOL CUP DMR HA and SYMBOL CUP DM CEM, a patient cohort with a minimum 2-year follow-up, 2-year follow-up data and sufficient numbers was only reached in 2018. The retrospective study proposed here is therefore the first clinical evaluation specific to these products.

The number of units of SYMBOL CUP DMR HA and SYMBOL CUP DM CEM fitted in France are summarized in Table 3 and Table 4 respectively.



Table 3: SYMBOL CUP DMR HA: Sales volume in France under this brand

| Year | 2014 | 2015 | 2016 | 2017 | Provisional<br>2018 |
|---|---|---|---|---|---|
| In public healthcare facilities | 0 | 0 | 4 | 8 | 16 |
| In non PHSPH private healthcare facilities | 15 | 194 | 98 | 128 | 155 |
| Total | 15 | 194 | 102 | 136 | 171 |

Table 4: SYMBOL CUP DM CEM: Sales volume in France under this brand

| Year | 2014 | 2015 | 2016 | 2017 | Provisional<br>2018 |
|---|---|---|---|---|---|
| In public healthcare facilities | 0 | 0 | 0 | 20 | 50 |
| In non PHSPH private healthcare facilities | 19 | 172 | 76 | 180 | 360 |
| Total | 19 | 172 | 76 | 200 | 410 |

The specific data resulting from this study will be used to establish the benefit-risk ratio of SYMBOL CUP DMR HA and SYMBOL CUP DM CEM. This information will enable:

- Update of the clinical evaluation for CE mark renewal purposes.
- An assessment of the product's application for inclusion in the Liste des Produits et Prestation Remboursables under the brand names by the Haute Autorité de Santé.

#### 2.3. STUDY HYPOTHESES AND EXPECTED RESULTS

The aim of this observational study is to estimate the risk and benefit of this implant in current clinical practice. As the approach is descriptive, no hypotheses have been made concerning the incidence of adverse events, or variations in endpoints during follow-up.

# 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. MAIN OBJECTIVE

Estimate the safety of these implants under normal conditions of use.



### 3.2. PRIMARY ENDPOINT

Implant survival rate at 2-year follow-up. This is the probability over time that the implant will remain in place in the living patient's hip. Events that reduce this probability are revision surgeries with removal of the implant, for whatever reason.

# 3.3. <u>SECONDARY OBJECTIVE</u>

Estimate the efficacy of these implants under normal conditions of use.

# 3.4. SECONDARY ENDPOINTS

- Safety: Intra and extra-prosthetic dislocation rates

- Safety: Incidence of other adverse events

- Effectiveness: Harris Hip Score (HHS)

- Effectiveness: Devane classification

Note: Since patients with no complaints requiring an orthopedic opinion do not usually present for a 2-year visit, only the functional questions of the 2-year HHS score will be collected during the telephone interview.

# 4. <u>DESCRIPTION OF THE STUDY</u>

The design of the study is:

- Observational
- Retrospective
- Non-comparative
- Not blinded
- Monocentric
- National

This methodologic choice is linked to the search of current practice data, and to the small number of surgeons who have so far use SYMBOL CUP DMR HA or SYMBOL CUP DM CEM, on large consecutive series of patients, thus enabling sufficient consecutive patient recruitment, and who, moreover, maintain a standard medical file record at 2-year follow-up with all the classic endpoints.

#### 4.1. DESCRIPTION OF MEASURES TAKEN TO REDUCE AND AVOID BIAS

Consecutive recruitment with provision of sampling frame data.



# 5. STUDY FEASABILITY

The clinical research associate (CRA) delegated by the sponsor will make two or three visits to the investigational center:

- An inclusion visit to confirm the investigator's adherence to the protocol and to define the procedures for extracting and transferring anonymized data from the electronic patient record management system. As this is a single-center study, this visit will take place before the protocol is submitted to the CNIL.
- A visit to extract and transfer anonymized data from patient files, and to call patients to obtain their two-year follow-up data. On this occasion, patients will be informed that they may object to the inclusion of their information in this study. During this visit, the sponsor's clinical research associate will check that the data are consistent with the contents of the patient files. He/she will confirm the completeness of the cohort, with consecutive placement of dual-mobility acetabular implants. An anonymized list of all THA during the recruitment period will be obtained and checked to establish the sampling frame. This visit will take place at the start of the study.
- An additional visit by the CRA, to obtain missing data and resolve discrepancies, will take place if necessary.

# 6. RÉALISATION PRATIQUE DU PROTOCOLE.

#### 6.1. <u>DEROULEMENT DES VISITES LIEES A L'ETUDE</u>

The clinical research associate (CRA) delegated by the sponsor will make two or three visits to the investigational center:

- An inclusion visit to confirm the investigator's adherence to the protocol and to define the procedures for extracting and transferring anonymized data from the electronic patient record management system. As this is a single-center study, this visit will take place before the protocol is submitted to the CNIL.
- A visit to extract and transfer anonymized data from patient files, and to call patients to obtain their two-year follow-up data. On this occasion, patients will be informed that they may object to the inclusion of their information in this study. During this visit, the sponsor's clinical research associate will check that the data are consistent with the contents of the patient files. He/she will confirm the completeness of the cohort, with consecutive placement of dual-mobility acetabular implants. An anonymized list of all THA during the recruitment period will be obtained and checked to establish the sampling frame. This visit will take place at the start of the study.



- An additional visit by the CRA, to obtain missing data and resolve discrepancies, will take place if necessary.

In the event of death reported by the patient's entourage without a date, the surgeon will question the civil registry of the patient's commune of birth to obtain the date and cause of death.

### **6.2. Summary of Patient Follow-up**

Patient follow-up is the surgeon's current practice. The protocol does not require any follow-up modalities additional to usual practice. In the event of missing data, the surgeon or secretariat will repeat a telephone call to the patients concerned, as usual, to ask follow-up questions. In the event of death reported by the patient's entourage without a date or explanation, the surgeon will question the civil registry of the patient's commune of birth.

# 6.3. DESCRIPTION OF THE GENERAL LOGISTICAL ORGANIZATION OF THE STUDY

The registered protocol and the copy of the database will be produced in 3 copies:

- The first to the investigator
- The second to the sponsor
- The third to the statistician.

All exchanges will be made by written mail transfer and USB key with acknowledgement of receipt. Any question raised by the statistician will be forwarded to the sponsor, who will obtain the investigator answer.

#### 6.4. BIOLOGICAL SAMPLES AND ANALYSES

Not applicable

## 7. ELIGIBILITY CRITERIA

## 7.1. <u>Inclusion criteria</u>

Any patient operated by Dr. Estour who has undergone hip replacement surgery with SYMBOL CUP DMR HA or SYMBOL CUP CEM acetabular implant and having reach 2-year follow-up on March 01, 2018.

#### 7.2. Non-inclusion criteria

Explicit refusal by the patient to allow data describing his pathology and treatment to be included in this study.

Minor patients or patients under guardianship.

# 7.3. RECRUITMENT PROCEDURES

As this study is retrospective, patients were recruiting during routine care prior to the drafting of protocol.

# 8. RULES FOR STOPPING THE STUDY

# 8.1. TERMINATION OF THE STUDY BY THE SPONSOR

The sponsor may stop the study at any time, for the following reasons:

- Major protocol violations,
- In the event of a request to stop by authorities

# 8.2. TERMINATION OF THE STUDY BY THE INVESTIGATOR

The investigator may stop participating in the study with agreement of the sponsor. The reason for the discontinuation of the study must be duly explained.

# 9. DATA COLLECTED

The data is collected in the electronic patient record management system will be copied directly into a spreadsheet by the surgeon or on site by the CRA. 2-year follow-up data will be entered directly into the spreadsheet. The list of variables is in Annex 2.

# 10. STATISTICAL CONSIDERATIONS

# 10.1. NUMBER OF SUBJECTS TO BE INCLUDED

The size of the cohort considered to be the minimum in light of studies carried out by other manufacturers is at least 20 with a follow-up of 2 years.

# 10.2. <u>Data analysis – General information: descriptive approach</u>

- Descriptive statistics: preoperative, operative, postoperative
- Tabulation of adverse events
- Kaplan-Meier analysis of implant survival
- Comparison tests of preoperative versus 1-year and 2-year postoperative efficacy scores.

Tests will be performed with a two-side alpha risk of 5%. Confidence intervals will be at 95%.

Continuous variables will be tested using Student's t-test. Categorial variables will be tested using Chi-2 test.



No subgroup analysis is planned.

No interim analysis is justified given the strict retrospective nature of the study.

# 10.3. MAIN ANALYSIS

Prothesis survival: Kaplan-Meier analysis.

# 10.4. SECONDARY ANALYSES

Subgroup analyses: Not applicable

- Descriptive statistics
- Continuous variables: Student's t-test or non-parametric tests in case of a breach of the conditions for applying parametric tests.
- Categorial variables: Chi-2 test.

# **10.5. SAMPLING FRAME**

The sampling frame, i.e. all patients operated by the same surgeon in the same institution, for total hip replacement, between the first and the last date of inclusion of patients in the SYMBOL CUP DMR HA or SYMBOL CUP DM CEM cohort, will be the subject of descriptive statistics.

Analysis will focus on age at date of operation, BMI, type of prosthesis, 1st intention or revision (See Questions relating to the sampling frame Annex 2).

Its characteristics will be compared to those of the cohort.

# 10.6. METHOD FOR TAKING INTO ACCOUNT MISSING, UNUSED OR INVALID DATA

As the statistical analysis is descriptive, it will be carried out « *per protocol* » and missing data will not be substituted by values derived from hypotheses.

Visibly aberrant data that the investigator cannot obtain through the usual telephone follow-up will be excluded from the analysis.

Adverse event or follow-up dates for which the day is missing will be substituted by the mid-month date.

# 10.7. PERSON RESPONSIBLE FOR THE ANALYSIS

DAOUD, Frédéric

Biostatistician

MEDEXTENS SARL

75 rue de Lourmel, 75015 Paris

Phone: 06 03 00 68 98

Mail: fcdaoud@medextens.com



Software used:

Data was analyzed in STATA 14.2 MP - Parallel Edition, 64-bit

StataCorp

4905 Lakeway Drive

College Station, Texas 77845 USA

2-core Stata perpetual license:

Serial number: 501406000407

Licence de Medextens SARL

### 11. ACCESS RIGHTS TO SOURCE DATA AND DOCUMENTS

#### 11.1. DATA ACCESS

The sponsor is responsible for obtaining the agreement of all parties involved in the study to guarantee direct access to all research sites, source data, source documents and reports for the purposes of quality control and audit by the sponsor.

Investigators will make available documents and individual data strictly necessary for the monitoring, quality control and auditing of biomedical research to persons with access to these documents in accordance with the legislative and regulatory provisions in force (articles L.1121-3 and R.5121-13 of the French Public Health Code).

#### 11.2. **SOURCE DATA**

Any original document or object that can be used to prove the existence or accuracy of a data item or fact recorded during the course of the research is defined as a source document.

The source data is exclusively the patient file located in the clinic where the patients included in the study were operated on, and under the responsibility of the surgeon.

The sponsor's CRA will be not able to obtain a copy of source data but may ask to check them to ensure the accuracy of the final database.

#### 11.3. DATA PRIVACY

In accordance with current legislation (articles L.1121-3 and R.5121-13 of the French Public Health Code), persons with direct access to source data must take all necessary precautions to ensure the confidentiality of information relating to investigational medicinal products, research, the persons



involved, and in particular their identity, as well as the results obtained. These persons, like the investigators themselves, are bound by professional confidentiality.

During biomedical research or at its termination, the data collected on the persons involved and transmitted to the sponsor by the doctors (or any other specialist) will be rendered anonymous. Under no circumstances may the names or addresses of the persons concerned should appear in clear text.

Patients will be coded by serial number. No initials will be recorded. Identification by the surgeon will be by month/year of birth, gender and date of surgery.

Source data form an integral part of the patient file.

The spreadsheet with extracted data sent to the sponsor wil be kept for 30 years after the medical device is withdrawn from the market.

The copy held by the statistician with the statistician scripts and data tables will be deleted by him from his company's computer as soon as the study report has been signed and submitted.

# 12. ETHICAL CONSIDERATIONS

# 12.1. INDEPENDENT ETHICS COMMITTEE

Not applicable

# **12.2.** PATIENT INFORMATION

Patients will be fully and fairly informed, in comprehensible terms, of the objectives of the study and the nature of the information collected, and of their right to object at any time to the use of the data collected. All this information is conveyed orally to patients by the surgeon. This oral information is completed by an information note given to each patient. Finally, general information on research activities is displayed at the Médipôle de Savoie Hospital.

# 12.3. SUPPORT FOR STUDY

This is a retrospective observational cohort study, whose only workload is the extraction of data from patient files. The cost of this work will be covered by the contract between the sponsor and the investigator once it has been approved by the CNOM.

# 13. DATA PROCESSING AND STORAGE OF DOCUMENTS AND DATA RELATING TO THE STUDY

# 13.1. DATA ENTRY AND PROCESSING

The data will be extracted into a spreadsheet by the investigator himself or his team in the institution. Analysis will be carried out by Frederic DAOUD See paragraph 10.7.

# 13.2. <u>CNIL</u>

This is a retrospective, single-center observational study. Thus, the study complies with the Reference Methodology MR003 and has been declared to the CNIL<sup>1</sup>.

# 13.3. ARCHIVING

The archiving of the documents mentioned below is the responsibility of DEDIENNE SANTE SAS. The documentation will be archived for a period of 30 years following withdrawal of the product from the market as defined in quality procedure PRO QUAL 001.

These documents are:

- Protocol et annexes, any amendments
- Information forms
- Database transferred by the investigator
- Follow-up documents
- Statistical report and any files used to produce the report
- Final study report

No displacement or destruction may be carried out without the agreement of the sponsor. At the end of the 30 years, the sponsor will be consulted for destruction. All data, documents and reports may be subject to audit or inspection.

# 14. COMMUNICATION – PUBLICATION RULES

Data will only be disclosed with the prior joint agreement of the investigator and the sponsor. The results may be communicated and published.

Website consulted:

https://www.legifrance.gouv.fr/affichTexte.do?cidTexte=JORFTEXT000033028290&dateTexte=&categorieLien=id

<sup>&</sup>lt;sup>1</sup> Official text: Deliberation no. 2016-263 of 21 July 2016 approving a reference methodology for the processing of personal data implemented in the context of research in the field of health that does not require the express or written consent of the data subject (MR-003).



# 15. INVESTIGATOR CONTRACT

See Annex 5

# 16. LIST OF ANNEXES

- Annex 1: Copy of CE mark and generic reimbursement code applicable to the patients included in the study
- Annex 2: List of study variables
- Annex 3: Information note and collection of non-opposition form
- Annex 4: CNIL registration
- Annex 5: Investigator contract

# 17. ASSOCIATED DOCUMENTS

Information note



# Annex 1: Copy of CE mark and generic reimbursement code applicable to the patients included in the study.

These products are currently supported under the following generic descriptions:

- SYMBOL CUP DM CEM: 3150450 hip, standard cup, modular, metal-back, without insert, cemented
- SYMBOL CUP DMR HA: 3168042 hip, reconstruction cup, modular, metal-back, without insert, uncemented
- DUAL MOBILITY PE LINER: 3161130 hip, solid polymer insert



ATTESTATION / CERTIFICATE N° 27262 rev. 5



Délivrée à Paris le 01 septembre 2015
Issued în Paris on September 1st, 2015

Certification Médical-Santé Notified Body N° 0459

# **ATTESTATION CE / EC CERTIFICATE**

Examen CE de la Conception (du produit) / EC Design Examination (of the product)
ANNEXE II point 4 de la directive 93/42/CEE relative aux dispositifs médicaux
ANNEX II section 4 DIRECTIVE 93/42/EEC concerning medical devices

Fabricant / Manufacturer

#### DEDIENNE SANTE

Le Mas des Cavaliers 217 rue Nungesser 34130 MAUGUIO FRANCE

Catégorie du(des) dispositif(s) / Device(s) category

Prothèse de l'articulation de la hanche - Cotyle double mobilité.

Hip joint prosthesis - Dual mobility cup.

Identification du(des) dispositif(s) / Identification of device(s)

SYMBOL CUP DM

(GMDN code 43167 - 43168)

See addendum

Le LNE/G-MED atteste qu'à l'examen des résultats figurant dans le(s) rapport(s) référencé(s) P122250 - P133684 - P137437 - P141487, le(s) produit(s) énuméré(s) ci-dessus est (sont) conforme(s) aux exigences de l'annexe I de la directive 93/42/CEE.

LNE/G-MED certifies that, on the basis of the results contained in the file(s) referenced P122250 - P133684 - P137437 - P141487, the product(s) complie(s) with the requirements of the directive 93/42/EEC, annex 1

Début de validité / Effective date : September 1st, 2015 (included) Valable jusqu'au / Expiry date : April 8th, 2019 (included)

On behalf of the Certification Director
Cécile VAUGELADE
G-MED Certification Division Manager

LNE - 27262 rev. 5 Modifie le certificat 27262-4

Laboratoire national de métrologie et d'essais • Établissement public à caractère industriel et commercial LNE/G-MED • Organisme notifié n° 0459

1, rue Gaston Boissier - 75724 Paris Cedex 15 • Tél.: 01 40 43 37 00 • Fax: 01 40 43 37 37 • www.lne.fr • www.gmed.fr

Page 22 sur 37





Addendum au certificat n° 27262 rev.5 page 1/2 Addendum of the certificate n° 27262 rev.5 Dossiers / Files N° P122250 - P133684 -P137437 - P141487

Certification Médical-Santé

# Identification des dispositifs / Identification of devices

| | Cotyle double mob<br>en chrome-coba<br>revêtu T | Cotyle double mobilité cimenté,<br>en chrome-cobalt (ISO 5832-4) | | | |
|---|---|---|---|---|---|
| SYMBOL CUP DM HA Metal-back standard, Ø 44 à Ø 68 | | SYMBOL CUP DMR HA Metal-back avec patte et trous pour plots, Ø 44 å Ø 68 | | SYMBOL CUP DM CEM<br>Metal-back standard, Ø 44 à Ø | |
| Taille 44 | 3700502203530 | Taille 44 | 3700502204087 | Taille 44 | 3700502203646 |
| Taille 46 | 3700502203547 | Taille 46 | 3700502204094 | Taille 46 | 3700502203653 |
| Taille 48 | 3700502203554 | Taille 48 | 3700502204100 | Taille 48 | 3700502203660 |
| Taille 50 | 3700502203561 | Taille 50 | 3700502204117 | Taille 50 | 3700502203677 |
| Taille 52 | 3700502203578 | Taille 52 | 3700502204124 | Taille 52 | 3700502203684 |
| Taille 54 | 3700502203585 | Taille 54 | 3700502204131 | Taille 54 | 3700502203691 |
| Taille 56 | 3700502203592 | Taille 56 | 3700502204148 | Taille 56 | 3700502203707 |
| Taille 58 | 3700502203608 | Taille 58 | 3700502204155 | Taille 58 | 3700502203714 |
| Taille 60 | 3700502203615 | Taille 60 | 3700502204162 | Taille 60 | 3700502203721 |
| Taille 62 | 3700502203622 | Taille 62 | 3700502204179 | Taille 62 | 3700502203738 |
| Taille 64 | 3700502203639 | Taille 64 | 3700502204186 | Taille 64 | 3700502203745 |
| Taille 66 | 3700502204957 | Taille 66 | 3700502204193 | Taille 66 | 3700502204971 |
| Taille 68 | 3700502204964 | Taille 68 | 3700502204209 | Taille 68 | 3700502204988 |

LNE/G-MED

0459



On behalf of the Certification Director Cécile VAUGELADE G-MED Certification Division Manager

ADD

720 DM 0701-31 rev 5 du 28/07/2015

Laboratoire national de métrologie et d'essais « Établissement public à caractère industriel et commercial LNE/G-MED » Organisme notifié n° 0459 |

1, rue Gaston Boissier - 75724 Paris Cedex 15 » TéL : 01 40 43 37 00 » Fax : 01 40 43 37 37 » www.lnc.fr » www.gmed fr





Certification Médical-Santé

Addendum au certificat nº 27262 rev.5

page 2/2

Addendum of the certificate n° 27262 rev.5 Dossiers / Files N° P122250 - P133684 -P137437 - P141487

| En UHMWPE (ISO 5834-2) pour cotyle dor<br>Insert pour tête Ø 22.2<br>Ø44 à Ø68 | | Insert pour tête Ø 28<br>Ø46 å Ø68 | |
|---|---|---|---|
| Taille 46 | 3700502203769 | Taille 46 | 3700502203868 |
| Taille 48 | 3700502203776 | Taille 48 | 3700502203875 |
| Taille 50 | 3700502203783 | Taille 50 | 3700502203882 |
| Taille 52 | 3700502203790 | Taille 52 | 3700502203899 |
| Taille 54 | 3700502203806 | Taille 54 | 3700502203905 |
| Taille 56 | 3700502203813 | Taille 56 | 3700502203912 |
| Taille 58 | 3700502203820 | Taille 58 | 3700502203929 |
| Taille 60 | 3700502203837 | Taille 60 | 3700502203936 |
| Taille 62 | 3700502203844 | Taille 62 | 3700502203943 |
| Taille 64 | 3700502203851 | Taille 64 | 3700502203950 |
| Taille 66 | 3700502203967 | Taille 66 | 3700502203981 |
| Taille 68 | 3700502203974 | Taille 68 | 3700502203998 |

LNE/G-MED

0459



On behalf of the Certification Director Cécile VAUGELADE G-MED Certification Division Manager

720 DM 0701-31 rev 5 du 28/07/2015

Laboratoire national de métrologie et d'essais « Établissement public à caractère industriel et commercial

LNEG-MED • Organisme notifié n° 0459 1. rue Gaston Boissier - 75724 Paris Cedex. 15 • Tél. : 01 40 43 37 00 • Fax : 01 40 43 37 37 • www.lne.fr • www.gmed.fr



# **Annex 2: List of study variables**

# DATA FROM THE COHORT SYMBOL CUP DMR HA AND SYMBOL CUP DM CEM

| PREOPERATIVE DEMOGRAPHICS | Order number of the surgery with this type of implant |
|---|---|
| | Type of implant DMR HA or CEM |
| | Month/year of birth |
| | Sex |
| | Surgeon identification |
| | Date of preoperative visit |
| | Height (cm) |
| | Weight (Kg) |
| | вмі |
| | BMI class |
| | Operated side |
| | Etiology / diagnosis |
| | Medication |
| | Medication - Specify |
| | Medical history |
| | Medical history - Specify |
| | Local surgical history on the affected hip |
| | Local surgical history on the affected hip - Specify |
| | Surgeon's comments |
| PREOPERATIVE | |
| DEVANE & CHARNLEY | |
| CLASSIFICATIONS | DEVANE |
| | CHARNLEY |
| HHS PAIN | Pain |
| HHS FUNCTIONAL ABILITIES -<br>WALKING | Lameness |
| WALKING | Support |
| | Walking perimeter |
| HHS FUNCTIONAL ABILITIES – | wanning perimeter |
| DAILY LIFE | Socks and shoes |
| | Stairs |
| | Sitting position |
| | Public transport |
| HHS – MOBILITY | Flexion ° |
| | Extension ° |
| | Abduction ° |
| | Adduction ° |
| | External rotation ° |



| | Internal rotation ° |
|---------------------------------|-------------------------------|
| | TOTAL MOBILITY |
| DEFORMATIONS | LLI (cm) |
| | Flessum ° |
| | Adductum ° |
| | Internal rotation ° |
| | TOTAL DEFORMATIONS |
| | TOTAL PREOPERATIVE HHS |
| SURGICAL INTERVENTION | Date of surgery |
| SONGICAL INTERVENTION | Age at surgery |
| | Intervention duration (min) |
| | Surgical approach |
| | Type of intervention |
| | Surgeon's comments |
| A CETA DALII A D. COMADONIENITO | Operative adverse events |
| ACETABULAR COMPONENTS | Cup walls |
| | Fragile acetabulum zone |
| | Cup identification |
| | Size |
| | Cement |
| | Reaming diameter |
| | Liner |
| | Femoral head |
| | Diameter |
| | Bone graft |
| | Screw |
| | Pegs |
| | Associated surgical procedure |
| FEMORAL STEM | Stem identification |
| | Cement |
| | CCD angle |
| | Collar |
| | Broach size |
| | Stem size |
| | Neck length |
| | Bone graft |
| STABILITY | Stability of the hip |
| INCIDENTS | Operative adverse events |
| SURGEON'S COMMENTS – END OF | aparatic describe cresses |
| SURGERY | Surgeon's comments |
| 1-year postoperative assessment | Date |
| | Death |



| | Reason for death |
|---|---|
| 1-year postoperative assessment | |
| DEVANE & CHARNLEY | |
| CLASSIFICATIONS | DEVANE |
| | CHARNLEY |
| HHS PAIN | Pain |
| HHS FUNCTIONAL ABILITIES - | |
| WALKING | Lameness |
| | Support |
| | Walking perimeter |
| HHS FUNCTIONAL ABILITIES – | |
| DAILY LIFE | Socks and shoes |
| | Stairs |
| | Sitting position |
| | Public transport |
| HHS – MOBILITY | Flexion ° |
| | Extension ° |
| | Abduction ° |
| | Adduction ° |
| | External rotation ° |
| | Internal rotation ° |
| | TOTAL MOBILITY |
| DEFORMATIONS | LLI (cm) |
| | Flessum ° |
| | Adductum ° |
| | Internal rotation ° |
| | TOTAL DEFORMATIONS |
| | TOTAL 1-YEAR FU HHS |
| Adverse events and reason | Adverse events at 1-year FU |
| | Date of occurrence of the adverse event |
| | Potential reason |
| Treatment | Without revision surgery |
| | Surgical revision without component revision |
| | Surgical revision with revision of components |
| | Date of revision surgery |
| | Adverse event solved Yes/No |
| | Unsolved adverse event – reason |
| Radiologic assessment at 1 year | Global offset |
| nadiologic assessment at 1 year | Global length |
| | Cup |
| | · |
| | Cup inclination |
| | Face stem |



| | Profile stem |
|---|---|
| | Surgeon's comments |
| 2-year postoperative assessment | Date of telephone interview |
| | Death |
| | Reason for death |
| 2-year postoperative assessment DEVANE & CHARNLEY | neason for death. |
| CLASSIFICATIONS | DEVANE |
| | CHARNLEY |
| HHS PAIN | Pain |
| HHS FUNCTIONAL ABILITIES - | |
| WALKING | Lameness |
| | Support |
| | Walking perimeter |
| HHS FUNCTIONAL ABILITIES – | |
| DAILY LIFE | Socks and shoes |
| | Stairs |
| | Sitting position |
| | Public transport |
| HHS FUNCTIONAL ABILITIES TOTAL | HHS FUNCTIONAL ABILITIES TOTAL AT 2-YEAR FU |
| Adverse events and reason | Adverse events at 2-year FU |
| | Date of occurrence of the adverse event |
| | Potential reason |
| Treatment | Without revision surgery |
| | Surgical revision without component revision |
| | Surgical revision with revision of components |
| | Date of revision surgery |
| | Adverse event solved Yes/No |
| | Unsolved adverse event – reason |



# SAMPLING FRAME DATA

| Patient number |
|---|
| Month/year of birth |
| Sex |
| Weight |
| Height |
| BMI |
| Date of surgery |
| Age at surgery |
| Type of intervention (first intention THA or revision THA) |
| Type of dual mobility acetabular implant (SYMBOL CUP DMR HA or SYMBOL CUP DM CEM) |
| Single or dual mobility |



#### **Annex 3. Information note**

#### Lettre d'information destinée au patient

# Etude de Cohorte Observationnelle Rétrospective SYMBOL CUP

Promoteur de l'étude : DEDIENNE SANTE SAS

Madame, Monsieur,

Vous avez bénéficié d'une chirurgie de prothèse totale de hanche avec un implant cotyloïdien à double-mobilité SYMBOL CUP DMR HA ou SYMBOL CUP DM CEM (fabriqué par la société DEDIENNE Santé) à l'Hôpital Médipôle de Savoie, avec le Dr. Gilles ESTOUR.

Le Dr. ESTOUR et la société DEDIENNE Santé réalisent actuellement la surveillance obligatoire des implants qui ont été posés. Pour cela nous examinons les détails de la chirurgie et du fonctionnement des implants au cours du temps sur l'ensemble des patients opérés entre mars 2015 et novembre 2016.

Cette note est destinée à vous donner des éléments d'informations sur l'étude clinique qui sera réalisée concernant cet implant. Si vous ne comprenez pas bien certains mots ou éléments de cette note, n'hésitez pas à demander des explications au médecin.

#### Présentation de l'étude

Cette étude sera menée dans le cadre d'une évaluation du niveau de sécurité et d'efficacité de cet implant dans des conditions habituelles d'utilisation. Il s'agit d'une recherche non interventionnelle : étude observationnelle, rétrospective, non comparative et monocentrique.

#### Objectifs de l'étude

L'objectif principal de l'étude est d'estimer le niveau de sécurité de l'implant dans des conditions habituelles d'utilisation, jusqu'à 2 ans post intervention chirurgicale.

Les objectifs secondaires de l'étude sont d'estimer l'efficacité de cet implant dans des conditions habituelles d'utilisation et jusqu'à 2 ans post intervention chirurgicale.

Cette étude permettra d'obtenir des données spécifiques au produit en question.

#### Méthodologie de l'étude

L'étude consiste en un recueil rétrospectif des données cliniques des sujets ayant bénéficié d'une mise en place d'une prothèse totale de hanche avec un implant cotyloïdien à double-mobilité SYMBOL CUP DMR HA ou SYMBOL CUP DM CEM :

- Issues des dossiers médicaux ou administratifs existants,
- Obtenues par interview téléphonique pour ce qui est des données jusqu'à 2 ans de suivi, si le dossier médical ne fournit pas toutes les informations sources.

# Contraintes et Obligations

Aucune contrainte et obligations.

Bénéfice potentiel attendu pour le participant et indemnisation

Il n'est pas attendu de bénéfice direct pour les personnes qui se prêtent à l'étude.

#### Risques engendrés du fait de la recherche

Il n'est pas attendu de risque lié à la participation à l'étude puisque l'intervention est réalisée dans un centre expert pour cette indication.

#### Droits et garanties des personnes

Dans le cadre de cette recherche, un traitement de vos données personnelles va être mis en œuvre afin de permettre l'analyse des résultats au regard de l'objectif de cette recherche. A cette fin, les données médicales vous concernant, identifiées par un numéro de code, seront transmises au promoteur. Elles pourront également, dans des conditions assurant leur confidentialité, être transmises aux autorités de santé françaises.



| Données Réglementaires Le protocole et le formulaire d'information seront soumis pour avis à la CNIL. La copie de l'enregistrement CNIL sera transmis au médecin coordonnateur. |
|---|
| Si vous avez des questions, n'hésitez pas à les poser au médecin. Dr Gilles ESTOUR |
| Chirurgien Orthopédiste Médipôle de Savoie 300 Avenue des Massettes 73190 Challes-les-Eaux Tél : 04 79 26 81 17 |
| Soyez assuré(e) que votre participation nous est extrêmement précieuse.<br>Nous vous remercions par avance, Madame, Monsieur de l'aide<br>que vous apportez ainsi à la recherche médicale. |



# **Annex 4. CNIL registration**



#### RÉCÉPISSÉ

### DÉCLARATION DE CONFORMITÉ À UNE MÉTHODOLOGIE DE RÉFÉRENCE

Numéro de déclaration

2176595 v 0

du 25 avril 2018

Monsieur TOLEDO Ludovic DEDIENNE SANTE DIRECTEUR GÉNÉRAL LE MAS DES CAVALIERS 217 RUE CHARLES NUNGESSER 34130 MAUGUIO

#### A LIRE IMPERATIVEMENT

La délivrance de ce récépissé atteste que vous avez transmis à la CNIL un dossier de déclaration formellement complet. Vous pouvez désormais mettre en œuvre votre traitement de données à caractère personnel.

La CNIL peut à tout moment verifier, par courrier, par la voie d'un contrôle sur place ou en ligne, que ce traitement respecte l'ensemble des dispositions de la loi, vous êtes tenu de respecter tout au long de votre traitement les obligations prévues et notamment :

- La définition et le respect de la finalité du traitement,
   La pertinence des données traitées,
- 3) La conservation pendant une durée limitée des données,
- 4) La sécurité et la confidentialité des données,
- 5) Le respect des droits des intéressés : information sur leur droit d'accès, de rectification et d'opposition.

Pour plus de détails sur les obligations prévues par la loi « informatique et libertés », consultez le site internet de la CNIL : www.cnil.fr.

# Organisme déclarant

Nom: DEDIENNE SANTE

Service:

Adresse: LE MAS DES CAVALIERS 217 RUE CHARLES

NUNGESSER

Code postal: 34130 Ville: MAUGUIO

N° SIREN ou SIRET:

339138638 00038

Code NAF ou APE:

3250A

Tél.: 0466280685 Fax.: 0466280692

Traitement déclaré

Finalité : MR3 - Recherches dans le domaine de la santé sans requeil du consentement

Transferts d'informations hors de l'Union européenne : Non

Fait à Paris, le 25 avril 2018 Par délégation de la commission

Isabelle FALQUE PIERROTIN Présidente



#### **Annex 5. Investigator contract**



#### PROJET DE CONVENTION

Selon article L.4113-6, loi Nº 2007-248 du 26 février 2007

- Préalablement à la présente convention, il est rappelé ce qui suit :
- " Est interdit le fait, pour les membres des professions médicales visées au titre 1er du livre IV du code de la santé publique, de recevoir des avantages en nature ou en espèces, sous quelque forme que ce soit, d'une façon directe ou indirecte, procurés par des entreprises assurant des prestations, produisant ou commercialisant des produits pris en charge par des régimes obligatoires de sécurité sociale.
- Toutefois, l'alinéa précédent ne s'applique pas aux avantages prévus par conventions passées entre les membres de ces professions médicales et des entreprises dès lors que ces conventions ont pour objet explicite et but réel des activités de recherche ou d'évaluation scientifique, qu'elles sont, avant leur mise en application, soumises pour avis au Conseil Départemental de l'Ordre des Médecins et notifiées lorsque les activités de recherche ou d'évaluation sont effectuées même partiellement, dans un établissement de santé, au responsable de l'établissement, et que les rémunérations ne sont pas calculées de manière proportionnelle au nombre de prestations ou produits prescrits, commercialisés ou assurés."

Extrait de l'article L4113-6 du code de la santé publique.

#### ENTRE:

1. La Société DEDIENNE SANTE, SAS au capital de 532 000 €, dont le siège social est à « Le Mas des Cavaliers » - 217, rue Nungesser - 34 130 Mauguio, inscrite au RCS de Montpellier sous le numéro 339 138 638, représentée par Ludovic TOLEDO, Directeur Général, ayant tous pouvoirs à l'effet des présentes,

Ft

2. Le Docteur Gilles ESTOUR (Identifiant RPPS : 10004039441), chirurgien orthopédiste exerçant à MEDIPOLE DE SAVOIE, Avenue des Massettes 73190 Challes-les-Eaux. et immatriculé à l'URSSAF en qualité de travailleur indépendant sous le n° 528 668 866, inscrit au Conseil Départemental de l'Ordre des Médecins de Savoie sous le numéro 73/3280.



#### ETANT PREALABLEMENT EXPOSE QUE:

Le Docteur Gilles ESTOUR développe une activité importante en chirurgie orthopédique, et que, dans ce domaine, il dispose de connaissances et d'un savoir-faire reconnus.

La Société DEDIENNE SANTE assure la fabrication et la distribution de prothèses et d'implants orthopédiques.

La Société DEDIENNE SANTE doit s'assurer de la qualité des résultats postopératoires obtenus avec les implants prothétiques qu'elle fabrique et distribue, notamment pour favoriser la valorisation technique et scientifique de ceux-ci, étant précisé que l'objet à court terme de cette convention est conforme à cet objectif.

Cette convention ne s'inscrit pas dans le cadre d'application de la loi HURIET, car il ne s'agit pas d'une expérimentation clinique prospective en vue de développer les connaissances biologiques et médicales mais de la validation d'un acte strictement thérapeutique. Elle répond aux critères d'une étude monocentrique puisqu'un seul centre a été chargé de suivre ce protocole.

#### IL EST CONVENU ET ARRETE CE QUI SUIT :

# ARTICLE 1: Mission

Le Docteur Gilles ESTOUR accepte de réaliser, pour le compte de la Société DEDIENNE SANTE, l'activité de suivi post-marché décrite ci-après :

- \* Produit(s) concerné(s): SYMBOL CUP DMR HA et SYMBOL CUP DM CIMENTE
- \* Nature des travaux. Recueil des informations objectives et quantifiées relatives à :
- la nature du diagnostic avant pose et l'indication retenue.
- le déroulement de l'intervention et le résultat opératoire obtenu.
- l'adéquation entre les tailles d'instruments et tailles d'instruments
- l'évolution postopératoire à 1 an et 2 ans, notamment du positionnement et du comportement de ces implants.

Il est entendu que le Docteur Gilles ESTOUR fera son possible pour assurer le suivi clinique de ses malades, afin que les résultats obtenus puissent être confirmés avec un plus grand recul clinique. Les informations seront consignées sur des cahiers d'observation spécifiques définis par la cellule d'évaluation clinique de la Société DEDIENNE SANTE, dont un exemplaire est joint à cette convention.

# Cadre de l'étude :

Dans le cadre de la directive 93/42/CEE, il s'agit d'assurer le suivi clinique postcommercialisation d'un dispositif médical marqué CE, afin de vérifier la sécurité et les performances revendiquées pour les dispositifs médicaux

Cette étude va permettre de collecter des données cliniques nécessaires à toute évolution des produits fabriqués par la Société DEDIENNE SANTE.



Ce suivi porte sur 20 dossiers de patients ayant un recul minimum de 2 ans. Les résultats correspondants seront transmis à la Société DEDIENNE SANTE. Il s'agit d'une étude rétrospective observationnelle.

Il est expressément mentionné que l'accomplissement de cette mission ne limite en rien l'indépendance du praticien et n'est assortie d'aucune obligation d'utilisation ou de prescription des produits de la Société DEDIENNE SANTE.

# ARTICLE 2 : Rémunération

Aucune rémunération au Docteur Gilles ESTOUR n'est prévue pour cette évaluation.

#### ARTICLE 3: Organisation

Pour favoriser la réalisation de ce suivi, DEDIENNE SANTE mettra à la disposition du Docteur les moyens informatiques nécessaires :

- Cahiers d'observation, ou fichier numérique.
- L'organisation et les moyens statistiques de la Cellule d'Evaluation Clinique de DEDIENNE SANTE.

#### ARTICLE 4: COMMUNICATION

La présente Convention sera communiquée pour avis par DEDIENNE SANTE au Conseil Départemental de l'Ordre des Médecins. Selon la loi du 2002-2013 du 4 mars 2002 relative aux droits des malades et à la qualité du système de santé, l'avis du Conseil de l'Ordre sera considéré comme favorable si un avis défavorable n'est pas transmis à DEDIENNE SANTE.

DEDIENNE SANTE transmettra au Docteur Gilles ESTOUR une copie de l'avis défavorable du Conseil de l'Ordre des Médecins, dans l'hypothèse de sa réception.

La présente Convention sera également portée, par le Docteur Gilles ESTOUR, à la connaissance du responsable de l'établissement dans les locaux duquel les travaux de suivi clinique seront opérés.

Les médecins hospitaliers ou hospitalo-universitaires, doivent en vertu du décret n° 2011-82 du 20 janvier 2011, obtenir l'autorisation du directeur de l'hôpital pour assurer une telle activité dite « accessoire ».

D'autre part, dans le souci de veiller au respect de la déontologie médicale les articles 4127-3 et 4127-5 du Code de la Santé Publique s'applique à cette Convention.

#### ARTICLE 5 : Confidentialité

Suivant l'article R5121-13 modifié par le Décret n°2012-597 du 27 avril 2012, les investigateurs et les personnes appelées à collaborer aux essais, sont tenus au secret professionnel en ce qui concerne notamment la nature des produits étudiés, les essais, les personnes qui s'y prêtent et les résultats obtenus.

Ils ne peuvent, sans l'accord du promoteur, donner d'informations relatives aux essais qu'au ministre chargé de la santé, aux médecins inspecteurs de santé publique, aux pharmaciens inspecteurs de santé publique, au directeur général et aux inspecteurs de l'ANSM.



Les essais ne peuvent faire l'objet d'aucun commentaire écrit ou oral sans l'accord conjoint de l'expérimentateur ou de l'investigateur et du promoteur.

#### ARTICLE 6: Validité

Il est entendu entre les parties que la validité de la présente convention est subordonnée à la réalisation par le Docteur Gilles ESTOUR et par la société DEDIENNE SANTE des obligations prévues dans le cadre de l'étude. Il est entendu en outre que la présente convention serait nulle et sans effet dans le cas où l'avis du Conseil de l'Ordre des Médecins serait défavorable.

#### ARTICLE 8

DEDIENNE SANTE se réserve le droit de publication des résultats observés.

Fait à Nîmes le 16/04/2018

en trois exemplaires :

1 exemplaire : DEDIENNE SANTE
 1 exemplaire : Docteur Gilles ESTOUR
 1 exemplaire pour le Conseil National de l'Ordre des Médecins

Docteur Gilles ESTOUR

Pour DEDIENNE SANTE M. Ludovic TOLEDO Directeur Général



# **18. BIBLIOGRAPHY**

<sup>1</sup> Avis de la CNEDIMTS du 18 novembre 2014 relatif à la phase contradictoire des prothèses de hanche. HAS, 2014.

ii Déclaration CE de conformité du 09 avril 2014.

iii Attestation CE – N°27262 rev. 5 du 1<sup>er</sup> septembre 2015. LNE, Organisme notifié n°0459. Cotyles Double mobilité sans ciment et à cimenter. SYMBOL CUP DM, GMDN code 43167-43168.

<sup>&</sup>lt;sup>iv</sup> Evaluation clinique «Cotyles de hanche, double mobilité, SYMBOL CUP DM » du 28/11/2013 réalisée par Dedienne Santé, mis à jour le 28/11/2014

VLNE G-MED. Revue et évaluation du rapport d'évaluation clinique. Evaluation initiale. DEDIENNE SANTE, DM: Cotyle double mobilité SYMBOL CUP DM, N° dossier: P122250. Rapport eval clinique DEDIENNE cotyle 2M SYMBOL 140214.pdf.